CLINICAL TRIAL: NCT02908932
Title: Ranger Resilience and Improved Performance on Phospholipid Bound Omega-3's
Acronym: RRIPP-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Aker BioMarine Human Ingredients AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00051532
Record Dates: First submitted 2016-08-24; First posted 2016-09-21 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Nutrition; Fatty Acids, Omega-3; Cognition; Resilience, Psychological; Psychology, Military

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phospholipid-bound omega-3 supplement (Experimental): 2.3g/d omega-3 HUFAs (with the EPA to DHA ratio of approximately 2:1), delivered in 8 capsules/day in Krill oil concentrates (Aker BioMarine Antarctic AS, Norway). Participants will receive supplements for the duration of IBOLC (19 weeks) and up until entry in Ranger. Time between completion of IBOLC and entry in Ranger is variable, ranging from 1 weeks to 10 weeks (4 weeks typical). Total duration on supplement thus ranges from 20 to 30 weeks.
  Interventions: Dietary Supplement: Phospholipid-bound omega-3 supplement
- Placebo supplement (Placebo Comparator): Matching placebo capsules, substituting macadamia nut oil and appropriate colorant for krill oil. Macadamia nut oil has not been associated with psychological, cognitive, or health benefits. Furthermore, it is not typically consumed in large quantities and is therefore useful in tracking blood serum levels to assess compliance within the placebo arm. Placebo capsules have been produced by Aker Biomarine. As with the experimental arm, participants will take 8 capsules daily for the duration of the study (20-30 weeks).
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Phospholipid-bound omega-3 supplement — The dietary supplement is produced by Aker BioMarine. These krill oil capsules received a GRAS status approval from the U.S. Food and Drug Administration (FDA) in 2010. Aker BioMarine has a new pending application (2015) with the U.S. FDA for GRAS status for its new product on which this study capsule is based. Aker BioMarine markets a number of different krill-based omega-3 supplement products in the U.S. The US Food and Drug Administration (FDA) has determined that an Investigator New Drug (IND) Application is not required for this study. This phospholipid-bound omega-3 dietary supplement is provided in capsule form.
  Arms: Phospholipid-bound omega-3 supplement
Dietary Supplement: Placebo supplement — Placebo capsules that are identical in size and color to the experimental but contain an equal amount of macadamia nut oil.
  Arms: Placebo supplement

SUMMARY:
The goal of this study is to determine if supplementation with krill oil concentrate containing the phospholipid-bound omega-3 fatty acids improves performance on specific cognitive tests that underlie key elements in U.S. Army Infantry Basic Officer Leaders Course (IBOLC) and in Ranger School (Training) at Fort Benning, Georgia (GA).

DETAILED DESCRIPTION:
The U.S. Army invests significant time and money in training its leaders. Individuals who choose the Army Infantry as their career expend significant time, energy, and commitment to self-development to achieve their career goals. While Infantry Basic Officer Leaders Course (IBOLC) graduates have demonstrated their ability to perform skills required for Ranger School success, personal stress during Ranger School appears to be a continual barrier to successful Ranger School graduation, with only 45.25% of IBOLC graduates having passed Ranger training in 2013. Omega-3 highly unsaturated fatty acids (HUFAs), specifically EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid), are concentrated in neural tissues, are essential for neural function (McNamara & Carlson, 2006 ), and must be obtained from dietary sources. United States (U.S.) food production practices over the last century have resulted in a dramatic change in the fatty acid profile of the U.S. diet. At the same time, evidence continues to build regarding the potential importance of omega-3 HUFAs on emotional state, cognitive function, and mental health. The purpose of this study is to investigate whether supplementation with omega-3 HUFAs from a krill oil concentrate will improve emotional status and related cognitive performance under stress among Infantry Officer Trainees during IBOLC, (Part I) and subsequent Ranger School (Part II). More broadly, Americans continue to report living under a high level of stress, with 20% reporting states of severe stress. The potential impact of this study would be information that would support the role for dietary supplementation of omega-3 HUFAs from krill oil concentrate in contributing to improving mood, emotional status, and cognitive performance among the U.S. population.

Overview: The Ranger Resilience and Improved Performance on Phospholipid Bound Omega-3's (RRIPP-3 Study) is a double-blinded, randomized, placebo-controlled trial conducted by the Medical University of South Carolina (MUSC) in partnership with the National Institutes of Health (NIH) working with the permission of the leadership of IBOLC and the U.S. Army Ranger Training School at Fort Benning, GA. Participants (450 individuals) will be randomized to one of two experimental groups for 2 Parts: Part I: IBOLC and Part II Ranger School.

Intervention Schedule: Participants will be provided with capsules of krill oil concentrate (2.3g/day HUFAs with EPA and DHA ratio of approximately 2:1) or placebo (macadamia nut oil and appropriate matching colorant for krill oil) delivered in 8 capsules per day during Part I (IBOLC training) only.

Compliance Monitoring: Finger prick blood samples will be collected for assessment of fatty acids at baseline and at specific time points during IBOLC and pre- and post-Ranger training and analyzed at a collaborating laboratory at the National Institutes of Health.

Study Participants: Sample Size: The sample size calculation is based on differences in one of the specific cognitive tests between the placebo and treatment groups based on prior omega-3 supplementation studies. The total sample size needed to detect the between groups difference is 352 (176 per group). Accounting for a potential attrition rate of 25%, the total number of enrolled subjects=450. Calculations were made using PASS 2008 software, (Version 08.0.13, Kaysvile, Utah).

Location, Population, and Recruitment Strategy: This study will be conducted at Fort Benning, GA with laboratory analytic support at NIH and MUSC. All healthy individuals who have arrived at Fort Benning to participate in IBOLC with the intention of continuing directly into Ranger Training after completion of IBOLC will be eligible for the study. Information about the RRIPP-3 Study will be available to IBOLC students upon arrival at Fort Benning prior to IBOLC. Those interested in potentially participating in the study can review the information about the study at the beginning of IBOLC and sign up for a screening/enrollment session. After seeing videos about the study and the informed consent process, and answering eligibility questions, if students remain interested, they will be asked to sign an informed consent and Health Insurance Portability and Accountability Act (HIPAA) for the baseline assessments. Once consent is obtained, the volunteer will participate in study baseline and enrollment, randomized, and provided with their omega-3 HUFA or placebo capsules.

Study Sessions: Overview: All participants will be expected to participate in 5 sessions held at Fort Benning. During the enrollment session a 24-hour dietary recall and 30-day food frequency questionnaire will be administered. Subsequent sessions will be scheduled at the 8 week check-in and two mid-points of IBOLC, and after leaving Ranger School (whether training is completed or not). Trained study coordinators will collect the data for the RRIPP-3 study. With the exception of the dietary assessment interview, the assessments for the RRIPP-3 study will be participant self-responses. Whether by self-response or coordinator interview, the responses will be collected directly into an automated, assessment order-sequenced computer test battery. With the exception of the informed consent documents, all participant information will be directly entered into the MUSC secure server as part of the RRIPP-3 study file. Participants will be assigned a study ID number at enrollment that will be used for the study duration. All data will be collected and filed in conjunction with the participant study identification (ID) number.

United States Department of Agriculture (USDA) Automated Multiple-Pass Method (AMPM) 24-Hour Dietary Assessment: AMPM (USDA, http://www.ars.usda.gov/Services/ ) is a computerized method for collecting interviewer-administered 24-hour dietary recalls in person. Food Frequency Questionnaire: The Diet History Questionnaire (DHQ) is a freely available food frequency questionnaire (FFQ). The DHQ II consists of 134 food items and 8 dietary supplement questions. RRIPP-3 will use the DHQ II electronic version which includes usual intake over the previous 30 days with portion size (NCI, 2010).

Data Coding and Analysis: Data will be collected and managed using REDCap electronic data capture tools hosted at MUSC (redcap.musc.edu) (Harris et al., 2009). All coded RRIPP-3 study data will be collected and separately transferred to the MUSC secure server. This coded data will be labeled only with the participant study id and participant randomization number. Adverse events will be reported using eIRB, South Carolina's federated online IRB system.

Randomization Scheme: The 2 treatment groups will be balanced with respect to commissioning source and post-graduation destination using a stratified blocked design.

Statistical Analysis Intent to treat and verified compliance assessments: All hypotheses will be tested using both "intent to treat" and "as-per-protocol" criteria.

Data Analysis: Improvement on critical facets of cognitive function during IBOLC (Part I) and Ranger School (Part II): Descriptive statistics (e.g. means, standard deviations, medians, percentages) will be used to characterize the 2 treatment groups. T-tests, chi-square tests, or non-parametric tests (Wilcoxon rank sum, Fisher's exact) will be used to compare baseline characteristics between groups. As IBOLC class unit may represent an intraclass correlation, a variable will be created to represent class representation in the combined model. In addition, time on intervention and time to Part II end-point may vary between subjects and thus may be adjusted for in analysis as appropriate.

The primary analyses will involve generalized linear mixed models (GLMMs) (with random subject effects) performed to determine whether group assignment to active or placebo treatment improves scores on cognitive function and psychological assessments. The primary outcomes measure for cognitive function from the cognitive and psychological measures are outlined above. Other intermediary variables will be included in the model as indicated. Hypothesis tests will be 2-tailed, and p-values will be compared to an overall alpha level of 0.05. Secondary analyses will be conducted to examine treatment efficacy in subject subgroups, although the statistical power may be lower for any such analyses given the reduced sample size. GLMMs and non-linear mixed models with random subject and intraclass cluster effects will be used as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Entry into IBOLC
2. No self-reported previous injuries that would impede potential physical performance success in IBOLC or Ranger training

Exclusion Criteria:

1. Infection, autoimmune disease, or fever of unknown origin
2. Coronary Heart Disease
3. History of seizures, except for febrile seizures during childhood
4. Known allergy to crustaceans (shellfish) or nuts
5. Vegetarian food preference.
6. Regular use of omega-3 containing supplements within the last 3 months.
7. Reported consumption of seafood three or more times per week within the last three months.
8. Carry diagnosis of Type I or Type II diabetes
9. Take hypoglycemic agents
10. Refusal to stop taking specific dietary supplements pertinent to the study with the exception of standard multivitamins during study participation
11. For women, pregnancy or intention to become pregnant during the potential study duration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change (vs. baseline) in Inhibition and Rule-Making | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Stroop
Change (vs. baseline) in psychological resiliency | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Connor-Davidson Resilience Scale (CD-RISC)
Group differences on Land Navigation scores (from IBOLC gradebook) | data collected by Army throughout 5 months of IBOLC training and scores summed at the end of 5 months and provided to study pi
  Land navigation tests the ability of candidates to navigate from one point to another using a map and compass while equipped with their individual combat gear.
Group differences on Marksmanship scores (from IBOLC gradebook) | data collected by Army throughout 5 months of IBOLC training and scores summed at the end of 5 months and provided to study pi
  The underlying construct, visual psychomotor control, is assessed by evaluating whether "Marksman" or higher ranking was achieved on first attempt.
Change (vs. baseline) in Focused Attention and Information processing speed | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Digit-Symbol Coding
Change (vs. baseline) in physiological resiliency | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Composite score from Patient Reported Outcomes Measurement Information System (PROMIS), v. 1.0 for Applied Cognition, Fatigue, & Sleep-related impairment

SECONDARY OUTCOMES:
Change (vs. baseline) in Working Memory | baseline, week 14, week 16,within 72 hours of ending Ranger training
  Figural Continuous Paired Associates Test (FCPAT; Turner, Drummond, Salamat, & Brown 2007)
Anxiety as a Measure of Psychological Functioning | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Anxiety: Spielberger State / Trait Anxiety Inventory (STAI; Speilberger 1983)
Stress Response | within 72 hours of ending Ranger training
  Peritraumatic Distress Inventory (PDI; Brunet et al. 2001)
Mood State as a measure of Psychological Functioning | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Mood State:Profile of Mood States - Bipolar (POMS-Bipolar;Lohr and McNair 1988)
Change (vs. baseline) in Reasoning | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Grammatical Reasoning (Lieberman, Caruso, Niro, & Bathalon 2006)
Change (vs. baseline) in Visual Attention | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Four-Choice Visual Reaction Time Test (Lieberman, Caruso, Niro, & Bathalon 2006)
Change (vs. baseline) in Decision-Making | baseline, week 14, week 16, within 72 hours of ending Ranger training
  Balloon Analogue Risk Task (BART: Lejuez et al., 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette P Marriott, PhD, Principal Investigator — Medical University of South Carolina; Travis H Turner, PhD, Principal Investigator — Medical University of South Carolina; Joseph R Hibbeln, MD, Principal Investigator — LMBB, NIAAA, NIH
Locations (3):
- United States (3):
  - US Army, Fort Benning, Fort Benning, Georgia
  - National Institutes of Health, Bethesda, Maryland
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antypa N, Smelt AH, Strengholt A, Van der Does AJ. Effects of omega-3 fatty acid supplementation on mood and emotional information processing in recovered depressed individuals. J Psychopharmacol. 2012 May;26(5):738-43. doi: 10.1177/0269881111424928. Epub 2011 Oct 16. PMID 22004690
- [Background] Antypa N, Van der Does AJ, Smelt AH, Rogers RD. Omega-3 fatty acids (fish-oil) and depression-related cognition in healthy volunteers. J Psychopharmacol. 2009 Sep;23(7):831-40. doi: 10.1177/0269881108092120. Epub 2008 Jun 26. PMID 18583436
- [Background] Blasbalg TL, Hibbeln JR, Ramsden CE, Majchrzak SF, Rawlings RR. Changes in consumption of omega-3 and omega-6 fatty acids in the United States during the 20th century. Am J Clin Nutr. 2011 May;93(5):950-62. doi: 10.3945/ajcn.110.006643. Epub 2011 Mar 2. PMID 21367944
- [Background] Appleton KM, Rogers PJ, Ness AR. Updated systematic review and meta-analysis of the effects of n-3 long-chain polyunsaturated fatty acids on depressed mood. Am J Clin Nutr. 2010 Mar;91(3):757-70. doi: 10.3945/ajcn.2009.28313. Epub 2010 Feb 3. PMID 20130098
- [Background] Bloch MH, Qawasmi A. Omega-3 fatty acid supplementation for the treatment of children with attention-deficit/hyperactivity disorder symptomatology: systematic review and meta-analysis. J Am Acad Child Adolesc Psychiatry. 2011 Oct;50(10):991-1000. doi: 10.1016/j.jaac.2011.06.008. Epub 2011 Aug 12. PMID 21961774
- [Background] Conklin SM, Harris JI, Manuck SB, Yao JK, Hibbeln JR, Muldoon MF. Serum omega-3 fatty acids are associated with variation in mood, personality and behavior in hypercholesterolemic community volunteers. Psychiatry Res. 2007 Jul 30;152(1):1-10. doi: 10.1016/j.psychres.2006.10.006. Epub 2007 Mar 23. PMID 17383013
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] de la Presa Owens S, Innis SM. Docosahexaenoic and arachidonic acid prevent a decrease in dopaminergic and serotoninergic neurotransmitters in frontal cortex caused by a linoleic and alpha-linolenic acid deficient diet in formula-fed piglets. J Nutr. 1999 Nov;129(11):2088-93. doi: 10.1093/jn/129.11.2088. PMID 10539789
- [Background] Dretsch MN, Johnston D, Bradley RS, MacRae H, Deuster PA, Harris WS. Effects of omega-3 fatty acid supplementation on neurocognitive functioning and mood in deployed U.S. soldiers: a pilot study. Mil Med. 2014 Apr;179(4):396-403. doi: 10.7205/MILMED-D-13-00395. PMID 24690964
- [Background] Fontani G, Corradeschi F, Felici A, Alfatti F, Migliorini S, Lodi L. Cognitive and physiological effects of Omega-3 polyunsaturated fatty acid supplementation in healthy subjects. Eur J Clin Invest. 2005 Nov;35(11):691-9. doi: 10.1111/j.1365-2362.2005.01570.x. PMID 16269019
- [Background] Freund-Levi Y, Eriksdotter-Jonhagen M, Cederholm T, Basun H, Faxen-Irving G, Garlind A, Vedin I, Vessby B, Wahlund LO, Palmblad J. Omega-3 fatty acid treatment in 174 patients with mild to moderate Alzheimer disease: OmegAD study: a randomized double-blind trial. Arch Neurol. 2006 Oct;63(10):1402-8. doi: 10.1001/archneur.63.10.1402. PMID 17030655
- [Background] Hallahan B, Hibbeln JR, Davis JM, Garland MR. Omega-3 fatty acid supplementation in patients with recurrent self-harm. Single-centre double-blind randomised controlled trial. Br J Psychiatry. 2007 Feb;190:118-22. doi: 10.1192/bjp.bp.106.022707. PMID 17267927
- [Background] Hibbeln JR. Fish consumption and major depression. Lancet. 1998 Apr 18;351(9110):1213. doi: 10.1016/S0140-6736(05)79168-6. No abstract available. PMID 9643729
- [Background] Hibbeln JR. Seafood consumption, the DHA content of mothers' milk and prevalence rates of postpartum depression: a cross-national, ecological analysis. J Affect Disord. 2002 May;69(1-3):15-29. doi: 10.1016/s0165-0327(01)00374-3. PMID 12103448
- [Background] Hibbeln JR, Gow RV. The potential for military diets to reduce depression, suicide, and impulsive aggression: a review of current evidence for omega-3 and omega-6 fatty acids. Mil Med. 2014 Nov;179(11 Suppl):117-28. doi: 10.7205/MILMED-D-14-00153. PMID 25373095
- [Background] Hibbeln JR, Linnoila M, Umhau JC, Rawlings R, George DT, Salem N Jr. Essential fatty acids predict metabolites of serotonin and dopamine in cerebrospinal fluid among healthy control subjects, and early- and late-onset alcoholics. Biol Psychiatry. 1998 Aug 15;44(4):235-42. doi: 10.1016/s0006-3223(98)00141-3. PMID 9715354
- [Background] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Glaser R. Omega-3 supplementation lowers inflammation and anxiety in medical students: a randomized controlled trial. Brain Behav Immun. 2011 Nov;25(8):1725-34. doi: 10.1016/j.bbi.2011.07.229. Epub 2011 Jul 19. PMID 21784145
- [Background] Kim HY, Spector AA, Xiong ZM. A synaptogenic amide N-docosahexaenoylethanolamide promotes hippocampal development. Prostaglandins Other Lipid Mediat. 2011 Nov;96(1-4):114-20. doi: 10.1016/j.prostaglandins.2011.07.002. Epub 2011 Jul 23. PMID 21810478
- [Background] Kotani S, Sakaguchi E, Warashina S, Matsukawa N, Ishikura Y, Kiso Y, Sakakibara M, Yoshimoto T, Guo J, Yamashima T. Dietary supplementation of arachidonic and docosahexaenoic acids improves cognitive dysfunction. Neurosci Res. 2006 Oct;56(2):159-64. doi: 10.1016/j.neures.2006.06.010. Epub 2006 Aug 14. PMID 16905216
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; AHA Nutrition Committee. American Heart Association. Omega-3 fatty acids and cardiovascular disease: new recommendations from the American Heart Association. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):151-2. doi: 10.1161/01.atv.0000057393.97337.ae. No abstract available. PMID 12588750
- [Background] Lavie CJ, Milani RV, Mehra MR, Ventura HO. Omega-3 polyunsaturated fatty acids and cardiovascular diseases. J Am Coll Cardiol. 2009 Aug 11;54(7):585-94. doi: 10.1016/j.jacc.2009.02.084. PMID 19660687
- [Background] Lieberman HR, Tharion WJ, Shukitt-Hale B, Speckman KL, Tulley R. Effects of caffeine, sleep loss, and stress on cognitive performance and mood during U.S. Navy SEAL training. Sea-Air-Land. Psychopharmacology (Berl). 2002 Nov;164(3):250-61. doi: 10.1007/s00213-002-1217-9. Epub 2002 Sep 5. PMID 12424548
- [Background] Lin YH, Hanson JA, Strandjord SE, Salem NM, Dretsch MN, Haub MD, Hibbeln JR. Fast transmethylation of total lipids in dried blood by microwave irradiation and its application to a population study. Lipids. 2014 Aug;49(8):839-51. doi: 10.1007/s11745-014-3918-3. Epub 2014 Jul 2. PMID 24986160
- [Background] Martins JG. EPA but not DHA appears to be responsible for the efficacy of omega-3 long chain polyunsaturated fatty acid supplementation in depression: evidence from a meta-analysis of randomized controlled trials. J Am Coll Nutr. 2009 Oct;28(5):525-42. doi: 10.1080/07315724.2009.10719785. PMID 20439549
- [Background] McNamara RK, Carlson SE. Role of omega-3 fatty acids in brain development and function: potential implications for the pathogenesis and prevention of psychopathology. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):329-49. doi: 10.1016/j.plefa.2006.07.010. Epub 2006 Sep 1. PMID 16949263
- [Background] McNamara RK, Able J, Jandacek R, Rider T, Tso P, Eliassen JC, Alfieri D, Weber W, Jarvis K, DelBello MP, Strakowski SM, Adler CM. Docosahexaenoic acid supplementation increases prefrontal cortex activation during sustained attention in healthy boys: a placebo-controlled, dose-ranging, functional magnetic resonance imaging study. Am J Clin Nutr. 2010 Apr;91(4):1060-7. doi: 10.3945/ajcn.2009.28549. Epub 2010 Feb 3. PMID 20130094
- [Background] Raskin R, Terry H. A principal-components analysis of the Narcissistic Personality Inventory and further evidence of its construct validity. J Pers Soc Psychol. 1988 May;54(5):890-902. doi: 10.1037//0022-3514.54.5.890. PMID 3379585
- [Background] Robinson JG, Ijioma N, Harris W. Omega-3 fatty acids and cognitive function in women. Womens Health (Lond). 2010 Jan;6(1):119-34. doi: 10.2217/whe.09.75. PMID 20088735
- [Background] Rogers PJ, Appleton KM, Kessler D, Peters TJ, Gunnell D, Hayward RC, Heatherley SV, Christian LM, McNaughton SA, Ness AR. No effect of n-3 long-chain polyunsaturated fatty acid (EPA and DHA) supplementation on depressed mood and cognitive function: a randomised controlled trial. Br J Nutr. 2008 Feb;99(2):421-31. doi: 10.1017/S0007114507801097. Epub 2007 Oct 24. PMID 17956647
- [Background] Salem N Jr, Litman B, Kim HY, Gawrisch K. Mechanisms of action of docosahexaenoic acid in the nervous system. Lipids. 2001 Sep;36(9):945-59. doi: 10.1007/s11745-001-0805-6. PMID 11724467
- [Background] Sublette ME, Hibbeln JR, Galfalvy H, Oquendo MA, Mann JJ. Omega-3 polyunsaturated essential fatty acid status as a predictor of future suicide risk. Am J Psychiatry. 2006 Jun;163(6):1100-2. doi: 10.1176/ajp.2006.163.6.1100. PMID 16741213
- [Background] Sublette ME, Milak MS, Hibbeln JR, Freed PJ, Oquendo MA, Malone KM, Parsey RV, Mann JJ. Plasma polyunsaturated fatty acids and regional cerebral glucose metabolism in major depression. Prostaglandins Leukot Essent Fatty Acids. 2009 Jan;80(1):57-64. doi: 10.1016/j.plefa.2008.11.004. Epub 2009 Jan 6. PMID 19128951
- [Derived] Turner TH, Newman JC, Marriott BP. Poor effort on cognitive testing in voluntary research predicts failure in US Army Ranger School: Implications for clinical trial design. Clin Trials. 2023 Dec;20(6):714-717. doi: 10.1177/17407745231178847. Epub 2023 Jun 2. PMID 37269077